CLINICAL TRIAL: NCT03312855
Title: Revacept, a Novel Inhibitor of Platelet Adhesion in Patients With Stable Coronary Artery Disease Undergoing Elective Percutaneous Coronary Interventions: a Phase II, Multicentre, Randomised, Double-blind and Placebo-controlled Study
Brief Title: Intracoronary Stenting and Antithrombotic Regimen: Lesion Platelet Adhesion as Selective Target of Endovenous Revacept
Acronym: ISAR-PLASTER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other); AdvanceCor GmbH (Industry); Technical University of Munich (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Revacept/CAD/02
Record Dates: First submitted 2017-10-13; First posted 2017-10-18 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Stable Coronary Artery Disease
Keywords: coronary artery disease; platelet inhibition
MeSH Terms: conditions — Coronary Artery Disease | interventions — Revacept

STUDY DESIGN:
Intervention Model Description: with 2 doses (80 and 160 mg) of Revacept versus placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Revacept 80 mg (Experimental): single dose, intravenous
  Interventions: Drug: Revacept 80 mg
- Revacept 160 mg (Experimental): single dose, intravenous
  Interventions: Drug: Revacept 160 mg
- Placebo (Placebo Comparator): single dose, intravenous
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Revacept 80 mg — single dose, intravenous application of 80 mg Revacept
  Arms: Revacept 80 mg
Drug: Revacept 160 mg — single dose, intravenous application of 180 mg Revacept
  Arms: Revacept 160 mg
Drug: Placebo — single dose, intravenous application of Placebo solution
  Arms: Placebo

SUMMARY:
The main objective is to evaluate the efficacy and safety of treatment with 2 doses (80 and 160 mg) of Revacept versus placebo in patients with stable coronary artery disease undergoing PCI.

DETAILED DESCRIPTION:
Revacept is a protein that is made up of an Fc fragment ("fragment crystallisable") fused to the GPVI receptor (the endogenous platelet collagen receptor). Consequently, Revacept binds to its ligand (collagen) on atherosclerotic plaques preventing circulating thrombocytes from binding to collagen exposed by the injured plaque. All this is achieved without affecting systemic hemostasis.

Thus, blocking of GPVI-dependent pathways by interfering with vascular collagen sites is commonly seen as an attractive target for an anti-platelet therapy of atherosclerotic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Men and women >18 years of age
* Diagnosis: Clinically stable coronary artery disease
* Angiographic evidence of coronary artery disease
* Indication for PCI

Exclusion Criteria:

* WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for up to 4 weeks after receiving investigational product.
* Women who are pregnant or breastfeeding or are planning pregnancy during course of trial
* Women with a positive pregnancy test on enrolment or prior to investigational product administration.
* Patients with elevated high sensitivity cardiac troponin T levels at screening
* Patients receiving antithrombotic therapy with Prasugrel or Ticagrelor within 7 days prior to randomisation
* History of hypersensitivity, contraindication or serious adverse reaction to any component of the study drug (GPVI-Fc, sucrose, mannitol), acetylsalicylic acid or clopidogrel
* History of bleeding diathesis or active bleeding within the last 30 days
* Recent intracerebral haemorrhage or trauma within the last 3 months
* Thrombocytopenia (platelet count <30000/mm3) at screening
* Sustained hypertension (systolic BP >179mmHg or diastolic BP >109mmHg) at screening
* Renal failure (estimated glomerular filtration rate < 30ml/min and/or dialysis)
* Severe systemic disease, such as known malignancies or other comorbid conditions with life expectancy less than one year that may result in protocol non-compliance
* Unable to provide informed consent (e.g. severe dementia, or psychosis)
* Current severe liver dysfunction (transaminase level >5-fold the upper normal range limit)
* Patients with an indication for anticoagulant therapy
* Participation in any other clinical interventional trial (drug/device) within less than 30 days prior to screening
* Any other contraindication to perform PCI
* Any planned additional PCI or surgery within 30 days after randomization
* Suspected poor capability to follow instructions and cooperate
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical illness (e.g. infectious disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
Primary endpoint-composite endpoint of death and myocardial injury | within 48 hours from randomisation
  A composite endpoint of death or myocardial injury (defined as increase in cardiac biomarker - high sensitivity cardiac troponin T of at least 5 times the upper limit of norm (ULN) within 48 hours from randomisation).

SECONDARY OUTCOMES:
All cause mortality | within 30 days after randomisation
  All cause mortality
Myocardial infarction | within 30 days after randomisation
  Myocardial infarction
PCI-related (type 4) myocardial infarction | within 30 days after randomisation
  PCI-related (type 4) myocardial infarction
Definite stent thrombosis | within 30 days after randomisation
  Definite stent thrombosis
Urgent coronary revascularization | within 30 days after randomisation
  Urgent coronary revascularization
Stroke | within 30 days after randomisation
  Stroke
Peak potprocedural high-sensitivity troponin T level | within 48 hours after randomisation
  Peak potprocedural high-sensitivity troponin T level
Bleeding class 2 or higher according to Bleeding Academic Research Consortium (BARC) criteria (safety endpoint) | within 30 days after randomisation
  Bleeding class 2 or higher according to Bleeding Academic Research Consortium (BARC) criteria (safety endpoint)

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Kastrati, MD, Study Chair — Deutsches Herzzentrum München; Steffen Massberg, MD, Study Chair — Klinikum der Universität München; Stefanie Schuepke, MD, Study Director — Deutsches Herzzentrum Muenchen
Locations (8):
- Germany (8):
  - Deutsches Herzzentrum München, Munich, Bavaria
  - Universitätsmedizin Berlin, Campus Benjamin Franklin, Berlin
  - Charité - Universitätsmedizin Berlin, Campus Virchow, Berlin
  - Universitätsklinikum Frankfurt, Medizinische Klinik III, Kardiologie, Frankfurt am Main
  - Universtätsmedizin Mainz, Zentrum für Kardiologie/Kardiologie I, Mainz
  - Klinikum der Universität München, Medizinische Klinik und Poliklinik I, Munich
  - Klinikum rechts der Isar, I. Medizinische Klinik und Poliklinik, Munich
  - Universitätsklinikum Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mayer K, Hein-Rothweiler R, Schupke S, Janisch M, Bernlochner I, Ndrepepa G, Sibbing D, Gori T, Borst O, Holdenrieder S, Kupka D, Petzold T, Bradaric C, Okrojek R, Leistner DM, Trippel TD, Munzel T, Landmesser U, Pieske B, Zeiher AM, Gawaz MP, Hapfelmeier A, Laugwitz KL, Schunkert H, Kastrati A, Massberg S. Efficacy and Safety of Revacept, a Novel Lesion-Directed Competitive Antagonist to Platelet Glycoprotein VI, in Patients Undergoing Elective Percutaneous Coronary Intervention for Stable Ischemic Heart Disease: The Randomized, Double-blind, Placebo-Controlled ISAR-PLASTER Phase 2 Trial. JAMA Cardiol. 2021 Jul 1;6(7):753-761. doi: 10.1001/jamacardio.2021.0475. PMID 33787834